CLINICAL TRIAL: NCT01821287
Title: Nutritional Failure in Infants With Single Ventricle Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-0638
Record Dates: First submitted 2013-03-11; First posted 2013-04-01 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Congenital Heart Disease; Nutritional Failure
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CHD Infants: Infants with a single ventricle (Congenital Heart Disease) CHD admitted to Cincinnati Children's Hospital Medical Center (CCHMC) for neonatal medical management or surgical palliation
  Interventions: Other: CHD
- Normal Controls: Healthy newborns (full-term infants with no known medical problems) recruited from Cincinnati Children's Hospital Medical Center (CCHMC) and private practices

INTERVENTIONS:
Other: CHD — The study is not providing an intervention but rather is observational/studying factors that could contribute to nutritional failure in single ventricle CHD infants
  Groups: CHD Infants

SUMMARY:
The purpose of this study is to understand the causes of growth failure and to define biochemical markers of nutritional failure in patients with single ventricle Congenital Heart Disease (CHD).

ELIGIBILITY:
Inclusion Criteria:

* CHD infants: Infants with a single ventricle CHD admitted to CCHMC for neonatal medical management or surgical palliation
* Normal controls: Healthy newborns (full-term infants with no known medical problems) recruited from CCHMC and private practices.

Exclusion Criteria:

* CHD infants: 1) Premature birth (<36 weeks), 2) Chromosomal abnormalities, 3) Major gastrointestinal, pulmonary or neurologic anomalies
* Normal controls: 1) Premature birth (<36 weeks), 2) Chromosomal abnormalities, 3) Major gastrointestinal, pulmonary or neurologic anomalies., 4) Cardiovascular anomalies

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants with Single Ventricle Congenital Heart Disease (CHD) being treated at CCHMC and Healthy newborns recruited from CCHMC and private practices
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Resting Energy Expenditure (REE) for infants with a single ventricle compared to the age-matched control infants using the analysis of covariance procedure | At 12 months of age
  The following covariates will be considered for inclusion in the model: cardiac diagnoses, measures of cardiac function, hemodynamic measurements, number of parents, and number of siblings living at home. Transformations of REE (e.g. log or rank) may be conducted to satisfy the assumptions of the analysis.

SECONDARY OUTCOMES:
The relationship between REE and weight changes in infants with a single ventricle and control subjects; measures include REE, weight, and z-score (weight for age) | At 12 months of age
  Will be estimated by Pearson's correlation coefficient. If the assumption of normality of the two measurements is not reasonable, Spearman's rank correlation will be conducted. To further explore the relationship between REE and weight gain in infants with a single ventricle, partial correlation coefficients will be estimated where the following covariates are considered for inclusion in the model: cardiac diagnoses, measures of cardiac function, number of parents, and number of siblings living at home.

OTHER OUTCOMES:
The relationship between biochemical markers of nutrition (prealbumin, IGF-1, IGFBP-3, IL6, IL8, TNF-α, cortisol, insulin, and lymphocyte subclasses) and weight changes in infants with a single ventricle | at newborn hospitalization (at 1-5 days)
  Will be estimated by Pearson's correlation coefficient. If the assumption of normality of the measurements is not reasonable, Spearman's rank correlation will be conducted. To further explore the relationship between biochemical markers of nutrition and weight gain, partial correlation coefficients will be estimated where the following covariates are considered for inclusion in the model: cardiac diagnoses, measures of cardiac function, number of parents, and number of siblings living at home. Finally, a regression model will be created using weight gain (and weight-for-age Z-scores) as the dependent variable and candidate independent variables including cardiac diagnoses, measures of cardiac function, hemodynamic measurements, REE, number of parents living at home, and number of siblings living at home

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Anderson, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States